CLINICAL TRIAL: NCT03350763
Title: Biliary Drainage Preceding Possible Pancreaticoduodenectomy. Are Self-expandable Metallic Stents (SEMS) Superior to Plastic Stents?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators busy with other projects at the moment
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, Head of department, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/2470/2017
Record Dates: First submitted 2017-11-18; First posted 2017-11-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Biliary decompression
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plastic biliary stent (Experimental): A plastic (ie Tannenbaum 10 Fr) biliary stent is used to achieve biliary decompression
  Interventions: Device: Tannenbaum 10 Fr biliary stent
- Self-expandable metallic biliary stent (Experimental): A self-expandable metallic biliary stent is used to achieve biliary decompression
  Interventions: Device: Self-expandable metallic biliary stent

INTERVENTIONS:
Device: Tannenbaum 10 Fr biliary stent — Tannenbaum 10 Fr biliary stent
  Arms: Plastic biliary stent
Device: Self-expandable metallic biliary stent — ie WallFlex biliary RX
  Arms: Self-expandable metallic biliary stent

SUMMARY:
This study looks in to the rate of biliary stent dysfunction for plastic and metallic stents in patients who need biliary drainage due to a tumor in pancreas before possible pancreaticoduodenectomy. Complications related to the biliary decompression, and possible post-surgical complications in all patients are also recorded.

This trial aims to confirm whether metallic biliary stents really are superior to plastic stents as some previous studies suggest. Specific patient groups are also evaluated individually to see, whether patients with ongoing cholangitis at the time of diagnosis or patients receiving neoadjuvant treatments have less stent dysfunction cases and complications with metallic stents than with plastic stents.

ELIGIBILITY:
Inclusion Criteria:

* Resectable tumor of the head of the pancreas
* Elevated serum bilirubin levels
* Radiologically visible dilatation of the biliary system

Exclusion Criteria:

* Distant metastasis
* Inoperable tumor or other reason, why the patient is unfit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stent failure rate, and need for re-procedure before pancreaticoduodenectomy. | Evaluation at the day of pancreatic surgery

SECONDARY OUTCOMES:
Other complications related to preoperative biliary decompression, and post-surgical complications | Complication emerged within 120 days from pancreaticoduodenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Leena Kylänpää, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Decker C, Christein JD, Phadnis MA, Wilcox CM, Varadarajulu S. Biliary metal stents are superior to plastic stents for preoperative biliary decompression in pancreatic cancer. Surg Endosc. 2011 Jul;25(7):2364-7. doi: 10.1007/s00464-010-1552-6. Epub 2011 Mar 4. PMID 21373939
- [Background] Haapamaki C, Seppanen H, Udd M, Juuti A, Halttunen J, Kiviluoto T, Siren J, Mustonen H, Kylanpaa L. Preoperative biliary decompression preceding pancreaticoduodenectomy with plastic or self-expandable metallic stent. Scand J Surg. 2015 Jun;104(2):79-85. doi: 10.1177/1457496914543975. Epub 2014 Jul 15. PMID 25028410
- [Background] Velanovich V, Kheibek T, Khan M. Relationship of postoperative complications from preoperative biliary stents after pancreaticoduodenectomy. A new cohort analysis and meta-analysis of modern studies. JOP. 2009 Jan 8;10(1):24-9. PMID 19129611